CLINICAL TRIAL: NCT04702074
Title: TCM Syndrome Differentiation Treatment on Reducing the Rehospitalization Rate of Discharged Elderly Patients With CAP:A Multi-center, Randomized, Double-blind Controlled Trial
Brief Title: TCM Syndrome Differentiation Treatment on Discharged Elderly Patients With CAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCM for discharged elderly CAP
Record Dates: First submitted 2021-01-01; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Community-acquired Pneumonia
Keywords: The discharged elderly patients with CAP; Syndrome differentiation of TCM; Randomized controlled trail
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese medicine granules (Experimental): The experimental group will be given Bu Fei Jian Pi Hua Tan granule or Yi Qi Yang Yin Qing Fei granule based on TCM syndrome differentiation.
  Interventions: Drug: Traditional Chinese medicine granules
- Traditional Chinese medicine granules placebo (Placebo Comparator): The control group will be given Bu Fei Jian Pi Hua Tan granule placebo or Yi Qi Yang Yin Qing Fei granule placebo based on TCM syndrome differentiation.
  Interventions: Drug: Traditional Chinese medicine granules placebo

INTERVENTIONS:
Drug: Traditional Chinese medicine granules — Bu Fei Jian Pi Hua Tan granule for syndrome of the lung and spleen qi deficiency and unclean phlegm dampness.
  Yi Qi Yang Yin Qing Fei granule for syndrome of qi and yin deficiency and unclean phlegm heat.
  Traditional Chinese medicine granules will be administered twice daily for 2 months.
  Arms: Traditional Chinese medicine granules
Drug: Traditional Chinese medicine granules placebo — Bu Fei Jian Pi Hua Tan granule placebo for syndrome of the lung and spleen qi deficiency and unclean phlegm dampness.
  Yi Qi Yang Yin Qing Fei granule placebo for Syndrome of qi and yin deficiency and unclean phlegm heat.
  Traditional Chinese medicine granules placebo will be administered twice daily for 2 months.
  The appearance, weight, color and odor of the preparation are the same as those of experimental group.
  The granule placebo consists of dextrin, bitter and 5% of the Traditional Chinese medicine granules .
  Arms: Traditional Chinese medicine granules placebo

SUMMARY:
This study is to evaluate the efficacy and safety of TCM syndrome differentiation treatment on the rehospitalization rate of discharged elderly patients with community acquired pneumonia(CAP)and to explore its mechanism.

DETAILED DESCRIPTION:
The incidence and mortality of elderly patients with CAP are on a rising trend, especially the mortality of those over 65 years old are the highest. The elderly patients with CAP have more complications and drug resistance, which makes it difficult to treat and have heavy burden on the society. The discharged elderly patients with CAP are still facing the risk of readmission or even death due to recurrent pneumonia or other reasons. Research reports showed that TCM syndrome differentiation treatment had a certain role in improving the condition of discharged elderly patients with CAP. Our previous exploratory studies suggested that TCM syndrome differentiation treatment on the discharged elderly patients with CAP had good clinical efficacy and safety.

This is a multi-center, randomized, double-blind, placebo controlled trial to evaluate the efficacy and safety of TCM syndrome differentiation on the rehospitalization rate of discharged elderly patients with CAP and to explore its mechanism. 292 patients will be randomly assigned in a 1:1 ratio to experimental group or control group for 2 months treatment and 6 months follow-up.The experimental group will be given by Bu Fei Jian Pi Hua Tan granule or Yi Qi Yang Yin Qing Fei granule based on TCM syndrome differentiation. The primary outcomes are rehospitalization rate. The secondary outcomes include mortality, assessment of disease severity(CURB65 scores),quality of life (SF-36), treatment satisfaction(ESQ-CAP),Clinician Reported Outcome for CAP,Patient Reported Outcome for CAP,nutritional status (MNA-SF).

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of discharged elderly patients with CAP within 1 weeks;
2. Syndrome differentiation meets criteria of syndrome of the lung and spleen qi deficiency and unclean phlegm dampness, Syndrome of qi and yin deficiency and unclean phlegm heat;
3. Age including or above 65 years old;
4. Voluntary treatment, oral medication;
5. With informed consent signed.

Exclusion Criteria:

1. A confirmed diagnosis of discharged elderly patients with severe CAP;
2. Patients with unconscious, dementia or mental disorders;
3. Patients with hydrothorax, bronchiectasis, active pulmonary tuberculosis, pulmonary abscess, chronic obstructive pulmonary disease of GOLD D;
4. Patients with aspiration risk of severe neuromuscular disorders and long-term bedridden;
5. Patients with tumor, severe cardiovascular disease and severe liver and kidney diseases;
6. Participants in clinical trials of other drugs;
7. People who are allergic to the treatment drugs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Rehospitalization rate | up to month 8.
  Rehospitalization and causes of rehospitalization during the study period will be recorded.

SECONDARY OUTCOMES:
Mortality | the month1,2 of treatment period and month3, 6 of follow-up period.
  Deaths and causes of death during the study period will be recorded.
CURB65 score | Before treatment, the month 2 of treatment period and month 6 of follow-up period.
  CURB65 score will be assessd the severity of discharged elderly patients with CAP. 0-1 points: in principle, outpatient treatment is enough; 2 points: hospitalization or out of hospital treatment under strict follow-up; 3-5 points: hospitalization. The higher scores will indicate the worse outcomes.
MNA-SF | Before treatment, the month 2 of treatment period and month 3, 6 of follow-up period.
  MNA-SF will be used to evaluate the nutritional status.The higher scores will indicate the better nutritional status.
CAP-PRO | Before treatment, the month 1,2 of treatment period and month 3, 6 of follow-up period.
  Patient Reported Outcome for CAP scale(CAP-PRO) will be used to evaluate clinical efficacy .The lower scores will indicate the better outcomes.
CAP-CRO | Before treatment, the month 1,2 of treatment period and month3, 6 of follow-up period.
  Clinician Reported Outcome for CAP scale(CAP-CRO)will be used to evaluate clinical efficacy . The lower scores will indicate the better outcomes.
SF-36 | Before treatment, the month 1,2 of treatment period and month 3, 6 of follow-up period.
  SF-36 will be used to evaluate quality of life with a total of 0-100. The higher scores will indicate the better quality of life.
ESQ-CAP | Before treatment, the month 1,2 of treatment period and month 3, 6 of follow-up period.
  The efficacy satisfaction questionnaire for CAP (ESQ-CAP) will be used to assess clinical efficacy. The higher scores will indicate the better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Henan University of Chinese Medicine, Zhengzhou, China